CLINICAL TRIAL: NCT00793442
Title: Endothelial Cell Signaling and Microcirculatory Flow in Severe Sepsis
Brief Title: Endothelium in Severe Sepsis
Status: Completed | Type: Observational
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Nathan Shapiro, Associate Professor of Emergency Medicine, Beth Israel Deaconess Medical Center
Other Study IDs: 2008P000089; 1R01HL091757-01A1 (NIH)
Record Dates: First submitted 2008-11-18; First posted 2008-11-19 (Estimated); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: Sepsis; Severe Sepsis; Septic Shock
Keywords: sepsis; severe sepsis; septic shock; endothelium; microcirculation; biomarkers
MeSH Terms: conditions — Sepsis; Shock, Septic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Novel Endothelial Markers Derivation: Our study participants will come from the Protocolized Care for Early Severe Sepsis (ProCESS) trial will be eligible participants.
  From the ProCESS subjects, the researchers will include those who were: 1) recruited by participating centers who participated in other components of this ancillary study or 2) who were sequentially enrolled from periods derived from the beginning, middle, and end of the ProCESS study.
  Interventions: Diagnostic Test: Blood Collection and Assays
- Novel Endothelial Marker Validation: Our study participants will come from the Protocolized Care for Early Severe Sepsis (ProCESS) trial will be eligible participants; the researchers will recruit a sequential 300 patient validation set.
  Interventions: Diagnostic Test: Blood Collection and Assays

INTERVENTIONS:
Diagnostic Test: Blood Collection and Assays — The researchers will sample blood upon enrollment, at 6 and 24 hours after the baseline sampling. The researchers will measure 6 different endothelial related biomarkers compromising different components of endothelial permeability and hemostasis.

SUMMARY:
The overall hypotheses of this project is that severe sepsis is associated with endothelial dysfunction; that endothelial dysfunction, in turn, is predictive of subsequent organ failure and death; and that protocolized resuscitation attenuates endothelial cell (EC) dysfunction and improves patient survival.

DETAILED DESCRIPTION:
The endothelial response is emerging as a critical element of sepsis pathophysiology. Preclinical data and small human studies suggest that endothelial cells are responsible for increased leukocyte adhesion, inflammation, activation of coagulation, and respond to increased levels of the endothelial cell mediator Vascular Endothelial Cell Growth Factor (VEGF). Furthermore, the endothelium plays an active role in microcirculatory homeostasis and the preservation of microvascular flow.

The researchers propose to study the endothelium by performing a comprehensive endothelial cell "read-out" through the measurement of circulating levels of endothelial cell biomarkers as well as direct visualization of microcirculatory flow with in-vivo videomicroscopy. Accordingly, the broad, long-term objective of this project is to study the role of the endothelium in sepsis in a large, heterogeneous group of patients. To accomplish this, the researchers will investigate two specific aims: 1) to study biomarkers of endothelial cell activation in sepsis; and, 2) to study microcirculatory flow in sepsis.

The overall hypotheses of this project is that severe sepsis is associated with endothelial dysfunction; that endothelial dysfunction, in turn, is predictive of subsequent organ failure and death; and that protocolized resuscitation attenuates endothelial cell (EC) dysfunction and improves patient survival. To test these hypotheses the researchers will utilize ancillary measurements (notably in-vivo assessment of microcirculatory flow), and additional samples and assays from the ProCESS clinical trial. ProCESS is a large, multicenter, randomized, controlled clinical trial testing the efficacy and mechanisms behind protocolized goal-directed resuscitation.

To conduct this line of investigation directed at the endothelium and microcirculation that was not addressed in the original trial, the researchers will select 8 ProCESS study sites for participation in this ancillary study. The researchers will directly visualize and quantify the presence of disturbances in sublingual microcirculatory flow utilizing the novel bedside technique of orthogonal polarization microscopy. Furthermore, the researchers will develop a multi-marker panel that assesses degree of endothelial cell dysfunction and subsequent mortality risk.

The researchers will also capitalize on the randomly assigned interventions in the ProCESS clinical trial to observe differences in endothelial response across the alternative resuscitation strategies. Improved understanding of these mechanisms may lead to strategies to predict outcome, to select patients for tailored (endothelium-directed) therapies, to follow treatment response, and to develop novel therapies for endothelial dysfunction in sepsis.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled as a participant in the ProCESS Trial (clinicaltrial.gov identifier NCT00510835)
* At least 18 years of age
* Suspected infection
* Two or more systemic inflammatory response syndrome (SIRS) criteria

  * Temperature </= 36˚ C or >/= 38˚C
  * Heart rate >/= 90 beats per minute
  * Mechanical ventilation for acute respiratory process or respiratory rate >/= 20 breaths per minute or PaC02 < 32 mmHg
  * WBC >/= 12,000/mm³ OR </= 4,000/mm³ OR > 10% bands
* Refractory hypotension (a systolic blood pressure < 90 mm Hg despite an IV fluid challenge of at least 20 ml/kg over a 30 minute period) or evidence of hypoperfusion (a blood lactate concentration >/= 4 mmol/L)

Exclusion Criteria:

* Known pregnancy
* Primary diagnosis of acute cerebral vascular event, acute coronary syndrome, -- acute pulmonary edema, status asthmaticus, major cardiac arrhythmia, active
* gastrointestinal hemorrhage, seizure, drug overdose, burn or trauma
* Requirement for immediate surgery
* ANC < 500/mm³
* CD4 < 50/mm³
* Do-not-resuscitate status
* Advanced directives restricting implementation of the protocol
* Contraindication to central venous catheterization
* Contradiction to blood transfusion (e.g., Jehovah's Witness)
* Treating physician deems aggressive care unsuitable
* Participation in another interventional study
* Transferred from another in-hospital setting
* inability to tolerate microscan procedure (eg oxygen requirement via face mack that can not be discontinue for the procedure)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Emergency department patients with severe sepsis
Sampling Method: Non-Probability Sample
Enrollment: 910 (Actual)
Dates: Start 2008-03 (Actual); Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Mortality | hospital mortality

SECONDARY OUTCOMES:
Organ Dysfunction assessed by Sepsis-related Organ Failure Assessment (SOFA) Score | first 72 hours

CONTACTS AND LOCATIONS:
Overall Officials: Nathan I Shapiro, MD, MPH, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (7):
- United States (7):
  - Universtiy of Alabama, Birmingham, Alabama
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - North Shore University Hospital, Manhasset, New York
  - Temple University Hospital, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - University of Utah Health Sciences Center, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hou PC, Filbin MR, Wang H, Ngo L, Huang DT, Aird WC, Yealy DM, Angus DC, Kellum JA, Shapiro NI; ProCESS Investigators( *). Endothelial Permeability and Hemostasis in Septic Shock: Results From the ProCESS Trial. Chest. 2017 Jul;152(1):22-31. doi: 10.1016/j.chest.2017.01.010. Epub 2017 Jan 19. PMID 28109962
- [Derived] Fabian-Jessing BK, Massey MJ, Filbin MR, Hou PC, Wang HE, Kirkegaard H, Yealy DM, Aird WC, Kellum JA, Angus DC, Shapiro NI; ProCESS Investigators. In vivo quantification of rolling and adhered leukocytes in human sepsis. Crit Care. 2018 Sep 30;22(1):240. doi: 10.1186/s13054-018-2173-z. PMID 30268146